CLINICAL TRIAL: NCT04282057
Title: Effect of an Aerobic Exercise Program Associated With Shock Wave Therapy Versus Radiofrequency on Skin and Subcutaneous Tissue: Randomized Controlled Study
Brief Title: Effects of Shockwave Therapy Versus Radiofrequency
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Escola Superior de Tecnologia da Saúde do Porto (Other)
Responsible Party: Principal Investigator, Andreia Noites, Teacher, Escola Superior de Tecnologia da Saúde do Porto
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AN-009
Record Dates: First submitted 2020-02-18; First posted 2020-02-24 (Actual); Last update posted 2020-09-30 (Actual); Status verified 2020-09

CONDITIONS: Cardiovascular Risk Factor; Metabolic Disease; Photoaging
Keywords: shock wave therapy; radiofrequency; adipose tissue; skin flaccidity; aerobic exercise
MeSH Terms: conditions — Metabolic Diseases | interventions — Extracorporeal Shockwave Therapy

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- shockwave therapy group (Experimental): This group performed aerobic exercise just after shock wave therapy in the abdominal region.
  Interventions: Device: Shock wave therapy
- radiofrequency group (Experimental): This group performed aerobic exercise just after radiofrequency in the abdominal region.
  Interventions: Device: Radiofrequency
- control group (Active Comparator): This group only performed aerobic exercise.
  Interventions: Device: Aerobic exercise

INTERVENTIONS:
Device: Radiofrequency — Radiofrequency protocol - The radiofrequency protocol was performed in dorsal decubitus, with the head elevated at 45 degrees. The application was in capacitive mode, with a 7cm electrode, always in movement. The duration of the application was established in 15 minutes, maintaining the local temperature between 40 to 42 celsius degrees at the epidermis.
  Arms: radiofrequency group
Device: Aerobic exercise — Aerobic exercise protocol - 40 minutes of aerobic moderate-intensity exercise (45-55% of reserve heart rate) using Karvonen's formula, performed on a cycloergometer. The duration of the exercise was divided into three parts: warm-up (5 minutes); body (30 minutes); and cooling (from 5 to 10 minutes). The entire protocol was monitored through the Polar® brand heart rate monitor and watch.
  Arms: control group
Device: Shock wave therapy — The shock wave device corresponds to the BTL-6000 X-Wave TM with a 20mm transmitter multifocal. The parameters used correspond to the pressure set between 2.8 and 3.5 bar, frequency 15 hertz and 3000 pulses per 10x15 cm area. It was used as a means contact gel for ultrasound, reference 033-051. In this procedure the participants found themselves in the supine position, with a pillow under the head and with the bending knees.
  Arms: shockwave therapy group

SUMMARY:
The main objective of this study is to compare the effect of 6 sessions of shock wave therapy versus radiofrequency followed by a protocol of moderate aerobic exercise, in the reduction of adiposity and abdominal flaccidity, in females between 18 and 60 years old. As a secondary objective, it is intended to understand the mechanism of fat mobilization by these two therapies.

DETAILED DESCRIPTION:
With the increasing awareness of the population regarding the high rate of obesity and the number of deaths per year as a result of being overweight, treatments for reducing measures are increasingly sought.

The evidence shows that the accumulation of fat located in the abdominal region is a risk factor for dyslipidemia and arterial hypertension, and a reduction in waist circumference can reduce the potential risk of cardiovascular disease.

In addition to this concern, with the aging of the population and changes in body dimensions due to pregnancy or to a weight loss process, body flaccidity is also a growing cosmetic complaint, and the result is a less firm and pending skin.

Physical exercise is a very important agent for combating excess weight, with special attention to aerobic physical exercise, which is able to decrease body fat tissue and increase the oxidation of fatty acids by 5 to 10 times more than in resting state. The evidence points out that the exercise prescription to decrease fat mass should focus on a high volume of training (30 to 60 minutes) with moderate intensity (40 to 60% of Heart Rate Reserve), performed regularly and mobilizing large muscle groups.

In order to combat abdominal adiposity, as well as the flaccidity of the region, radiofrequency is presented as a possible complementary strategy.

Radiofrequency is an electromagnetic wave that when applied to skin, generates oscillating magnetic fields that move electrically charged particles producing heat in the tissues. The amount of heat produced is dependent on resistance.

Shock wave therapy consists of the application of high energy acoustic waves whose main characteristic is the production of a high pressure pulse induced in a short period of time. This will generate mechanical pressure waves in the tissues, promoting cavitation, with the formation of gas bubbles in the intervening fluids and an increase in local temperature.

The main objective of this study is to compare the effect of 6 sessions of shock wave therapy versus radiofrequency followed by a protocol of moderate aerobic exercise, in the reduction of adiposity and abdominal flaccidity, in females between 18 and 60 years old. As a secondary objective, it is intended to understand the mechanism of fat mobilization by these two therapies.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 18 to 60 years

Exclusion Criteria:

* smoking and drinking habits;
* athletes;
* people with dietary restrictions;
* participants who have had diets to lose weight in the last 3 months or who will start during the study;
* pregnant women;
* in postpartum less than one year;
* breastfeeding;
* intending to become pregnant during the study period;
* patients with electronic or metallic devices (pacemaker, IUD);
* individuals with metabolic (including dyslipidemias);
* hematological and renal disorders;
* individuals with dermatological changes;
* cardiovascular, respiratory, digestive, orthopedic, rheumatological and oncological pathologies;
* changes in the immune system or with acute inflammatory processes;
* changes in sensitivity or subject to medication (anti-coagulants, corticosteroids up to 6 weeks before, non-steroidal anti-inflammatory drugs, antihistamines, diuretics)

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2020-02-22 (Actual); Primary Completion 2020-04-25 (Actual); Study Completion 2020-06-19 (Actual)

PRIMARY OUTCOMES:
Cutaneous abdominal tissue thickness | Baseline
  Measurement of the cutaneous fold by ultrasonography
Cutaneous abdominal tissue thickness | 3 weeks after
  Measurement of the cutaneous fold by ultrasonography
Cutaneous abdominal tissue thickness | 6 weeks after
  Measurement of the cutaneous fold by ultrasonography
Subcutaneous abdominal tissue thickness | Baseline
  Measurement of the subcutaneous adipose fold by ultrasonography
Subcutaneous abdominal tissue thickness | 3 weeks after
  Measurement of the subcutaneous adipose fold by ultrasonography
Subcutaneous abdominal tissue thickness | 6 weeks after
  Measurement of the subcutaneous adipose fold by ultrasonography
Glycerol concentration | Baseline
  Blood analysis collection carried out with help from an clinical analysis technician
Glycerol concentration | 3 weeks after
  Blood analysis collection carried out with help from an clinical analysis technician
Glycerol concentration | 6 weeks after
  Blood analysis collection carried out with help from an clinical analysis technician
Lipid profile (LDL, HDL and triglyceride concentrations) | Baseline
  Blood analysis collection carried out with help from an clinical analysis technician
Lipid profile (LDL, HDL and triglyceride concentrations) | 3 weeks after
  Blood analysis collection carried out with help from an clinical analysis technician
Lipid profile (LDL, HDL and triglyceride concentrations) | 6 weeks after
  Blood analysis collection carried out with help from an clinical analysis technician
Perimetry | Baseline
  Perimetry consists of measuring circumferences. In this case, of the waist at the navel area, 3 cm below it and in the hip area
Perimetry | 3 weeks after
  Perimetry consists of measuring circumferences. In this case, of the waist at the navel area, 3 cm below it and in the hip area
Perimetry | 6 weeks after
  Perimetry consists of measuring circumferences. In this case, of the waist at the navel area, 3 cm below it and in the hip area
Adipometry | Baseline
  Adipometry consists of measuring skinfold thickness
Adipometry | 3 weeks after
  Adipometry consists of measuring skinfold thickness
Adipometry | 6 weeks after
  Adipometry consists of measuring skinfold thickness
Inflammatory markers concentration (IL6, CRP, TNF) | Baseline
  Blood analysis collection carried out with help from an clinical analysis technician
Inflammatory markers concentration (IL6, CRP, TNF) | 3 weeks after
  Blood analysis collection carried out with help from an clinical analysis technician
Inflammatory markers concentration (IL6, CRP, TNF) | 6 weeks after
  Blood analysis collection carried out with help from an clinical analysis technician
Nitrous oxide concentration | Baseline
  Blood analysis collection carried out with help from an clinical analysis technician
Nitrous oxide concentration | 3 weeks after
  Blood analysis collection carried out with help from an clinical analysis technician
Nitrous oxide concentration | 6 weeks after
  Blood analysis collection carried out with help from an clinical analysis technician
Body composition- body mass | Baseline
  body mass in kilograms
Body composition- body mass | 3 weeks after
  body mass in kilograms
Body composition- body mass | 6 weeks after
  body mass in kilograms
Body composition- muscle mass | Baseline
  muscle mass in kilograms
Body composition- muscle mass | 3 weeks after
  muscle mass in kilograms
Body composition- muscle mass | 6 weeks after
  muscle mass in kilograms
Body composition- fat mass | Baseline
  fat mass in kilograms
Body composition- fat mass | 3 weeks after
  fat mass in kilograms
Body composition- fat mass | 6 weeks after
  fat mass in kilograms
Body composition- visceral fat | Baseline
  visceral fat
Body composition- visceral fat | 3 weeks after
  visceral fat
Body composition- visceral fat | 6 weeks after
  visceral fat
Body composition- fat body areas | Baseline
  percentage of fat distributed by body areas
Body composition- fat body areas | 3 weeks after
  percentage of fat distributed by body areas
Body composition- fat body areas | 6 weeks after
  percentage of fat distributed by body areas
Thermography | Baseline
  Thermography is used to assess the temperature of the skin surface, and it is also possible to suppose changes in blood flow and vascularization with this outcome
Thermography | 3 weeks after
  Thermography is used to assess the temperature of the skin surface, and it is also possible to suppose changes in blood flow and vascularization with this outcome
Thermography | 6 weeks after
  Thermography is used to assess the temperature of the skin surface, and it is also possible to suppose changes in blood flow and vascularization with this outcome
Photography | Baseline
  Photography is used to compare the before and after images. With these it is possible to evaluate the skin flaccidity and fat
Photography | 3 weeks after
  Photography is used to compare the before and after images. With these it is possible to evaluate the skin flaccidity and fat
Photography | 6 weeks after
  Photography is used to compare the before and after images. With these it is possible to evaluate the skin flaccidity and fat

SECONDARY OUTCOMES:
skin flaccidity | Baseline
  Investigator Assessment Skin Laxity Scoring System - Questionnaire that evaluates skin flaccidity and scores from 0 to 4. (As the subjectivity assessment of this outcome, the investigator who evaluates is blind to the group that the participants are allocated, in order to avoid partial scores)
skin flaccidity | 3 weeks after
  Investigator Assessment Skin Laxity Scoring System - Questionnaire that evaluates skin flaccidity and scores from 0 to 4. (As the subjectivity assessment of this outcome, the investigator who evaluates is blind to the group that the participants are allocated, in order to avoid partial scores)
skin flaccidity | 6 weeks after
  Investigator Assessment Skin Laxity Scoring System - Questionnaire that evaluates skin flaccidity and scores from 0 to 4. (As the subjectivity assessment of this outcome, the investigator who evaluates is blind to the group that the participants are allocated, in order to avoid partial scores)
skin flaccidity and localized fat in the abdomen region | Baseline
  Satisfaction questionnaire to evaluate the final results according to the participant
skin flaccidity and localized fat in the abdomen region | 3 weeks after
  Satisfaction questionnaire to evaluate the final results according to the participant
skin flaccidity and localized fat in the abdomen region | 6 weeks after
  Satisfaction questionnaire to evaluate the final results according to the participant

CONTACTS AND LOCATIONS:
Locations (1):
- Andreia Noites, Vila Nova de Gaia, Porto District, Portugal

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Adatto MA, Adatto-Neilson R, Novak P, Krotz A, Haller G. Body shaping with acoustic wave therapy AWT((R))/EPAT((R)): randomized, controlled study on 14 subjects. J Cosmet Laser Ther. 2011 Dec;13(6):291-6. doi: 10.3109/14764172.2011.630089. PMID 21981441
- [Background] Modena DAO, da Silva CN, Grecco C, Guidi RM, Moreira RG, Coelho AA, Sant'Ana E, de Souza JR. Extracorporeal shockwave: mechanisms of action and physiological aspects for cellulite, body shaping, and localized fat-Systematic review. J Cosmet Laser Ther. 2017 Oct;19(6):314-319. doi: 10.1080/14764172.2017.1334928. Epub 2017 Jun 7. PMID 28590827
- [Background] Noites A, Vale AL, Pereira AS, Morais A, Vilarinho R, Carvalho P, Amorim M, Moreira T, Mendonca A. Effect of an aerobic exercise session combined with abdominal radiofrequency on lipolytic activity in women: Randomized control trial. J Cosmet Dermatol. 2020 Mar;19(3):638-645. doi: 10.1111/jocd.13056. Epub 2019 Jun 29. PMID 31254455
- [Background] Vale AL, Pereira AS, Morais A, de Carvalho P, Vilarinho R, Mendonca A, Noites A. Effect of four sessions of aerobic exercise with abdominal radiofrequency in adipose tissue in healthy women: Randomized control trial. J Cosmet Dermatol. 2020 Feb;19(2):359-367. doi: 10.1111/jocd.13036. Epub 2019 Jun 3. PMID 31157522